CLINICAL TRIAL: NCT04053894
Title: Association of PeriOPerative Aspirin-ResisTance and CardioVascular Outcome
Acronym: POPART-CVO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Jan Larmann, Attending Anesthesiologist, University Hospital Heidelberg
Other Study IDs: S-468/2019
Record Dates: First submitted 2019-08-09; First posted 2019-08-13 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Vascular Surgery
Keywords: vascular surgery; aspirin resistance; MINS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of our study is to investigate the association between perioperative aspirin resistance and Myocardial Injury after Non-cardiac Surgery (MINS) in patients undergoing vascular surgery.

DETAILED DESCRIPTION:
Because of new surgical techniques, advanced monitoring modalities and improvements in perioperative care, perioperative mortality and morbidity have been significantly reduced in the last decades; however, patients still suffer from high perioperative mortality and morbidity, especially those with pre-existing cardiovascular diseases. Not only perioperative myocardial infarction but also myocardial injury after non-cardiac surgery, which presents without clinical symptoms, is associated with an adverse outcome. Possibilities to preoperatively identify patients at cardiovascular risk are limited and prophylactic interventions are not yet established or controversial.

Aspirin is used for primary and secondary prevention in cardiovascular diseases. New-onset increased platelet function on aspirin treatment (aspirin resistance) has been demonstrated in cardiac and vascular surgery. Yet, it has not been investigated whether a new perioperative aspirin resistance is associated with higher risk of myocardial injury after non-cardiac surgery (MINS) and cardiovascular events.

The aim of this study is to evaluate a potential association between new-onset aspirin resistance and MINS in patients undergoing vascular surgery. If there is an association of perioperative aspirin resistance and MINS during vascular surgery, the detection of perioperative aspirin resistance could be used as perioperative risk stratification tool in order to improve clinical risk stratification and reduce perioperative morbidity and mortality.

Therefore, 220 patients treated with aspirin and scheduled for vascular surgery will be recruited. Blood will be drawn at predefined time points before surgery and up to three days postoperatively. Aspirin resistance will be measured by Multiplate Analyzer prior to surgery, one hour after skin-incision, four hours after surgery and on post-OP days one and two. Adverse cardiovascular events will be recorded until 30 days post-OP. ECGs will be recorded preoperatively and on post-OP day 3. High-sensitive cardiac Troponin T will be measured prior to surgery and on post-OP days one to three. Patient charts will be screened and a telephone interview will be performed to detect cardiovascular events after discharge until post-OP day 30.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Preoperative aspirin treatment at least 14 days prior to surgery
* Elective vascular surgery
* In-patient treatment
* Informed consent

Exclusion Criteria:

* 17 years of age or younger
* Known pregnancy or breastfeeding
* Missing informed consent
* Ambulatory or day-case surgery
* Emergency surgery
* Current clopidogrel or non-steroidal anti-inflammatory drug treatment
* Preoperative aspirin resistance
* Current thrombocytopenia (<100000 platelet/µl)
* Liver or renal failure (GOT/GPT and/or creatinine increased >2-fold)
* Entity which is part of the composite endpoint diagnosed within past 28 days
* Angiography without surgical intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients on aspirin treatment, admitted to University Hospital Heidelberg and scheduled for vascular surgery.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Myocardial Injury after Non-cardiac Surgery | 30 days postoperative
  Number of participants with MINS defined as raise in postoperative hs-cTNT (high sensitivity cardiac troponin T) judged due to myocardial ischemia detected at postoperative visits, documented in patient chart or detected during telephone interview after 30 postoperative days.

SECONDARY OUTCOMES:
Composite of Cardiovascular Events | 30 days postoperative
  Number of participants with Cardiovascular Events defined as occurrence of Cardiac Death and/or Myocardial Ischemia and/or Myocardial Infarction and/or Embolic Stroke and/or Thrombotic Stroke recorded until postoperative day 30. Definitions according to European Perioperative Clinical Outcome-(EPCO) detected at postoperative visits, documented in patient chart or detected during telephone interview after 30 postoperative days
Peripheral vascular occlusion | 30 days postoperative
  Diagnosed by a radiologist based on the results of duplex ultrasonography, angiography or CT-angiography.
Mesenteric ischemia | 30 days postoperative
  Diagnosed by a radiologist based on the results of angiography or CT-angiography.
New-onset atrial fibrillation | 30 days postoperative
  Number of participants with new electrocardiographic detection of atrial fibrillation in postoperative ECG and/or documented in patient chart
Congestive heart failure | 30 days postoperative
  Number of participants with congestive heart failure according to European Perioperative Clinical Outcome (EPCO) definitions
Cardiac death | 30 days postoperative
  Number of participants with cardiac death defined as death due to new myocardial infarction or ischemia, or atrial or ventricular arrhythmias, or cardiogenic pulmonary edema, or pulmonary embolism detected at postoperative visits, documented in patient chart or detected during telephone interview after 30 postoperative days
Myocardial Ischemia | 30 days postoperative
  Number of participants with myocardial ischemia defined as new electrocardiographic detection of myocardial ischemia in ECG and/or documented in patient charts which will be screened up to 30 postoperative days and/or detected during telephone interview after 30 postoperative days
Myocardial Infarction | 30 days postoperative
  Number of participants with myocardial infarction defined as an increase in serum cardiac biomarker values in combination with symptoms of ischemia or new/presumed new significant ST segment or T wave ECG changes or new left bundle branch block or development of pathological Q waves on ECG. Definition according to European Perioperative Clinical Outcome-(EPCO) detected at postoperative visits, postoperative blood analyses, documented in patient chart or detected during telephone interview after 30 postoperative days
Stroke | 30 days postoperative
  Number of participants with embolic or thrombotic stroke defined as cerebral event with persistent residual motor, sensory or cognitive dysfunction detected at postoperative visits, documented in patient chart or detected during telephone interview after 30 postoperative days.
Length of hospital stay | 30 days postoperative
  Documented in patient charts.
Length of intensive care unit stay | 30 days postoperative
  Documented in patient charts.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Larmann, MD PhD, Principal Investigator — Departement of Anaesthesiology, Heidelberg University Hospital
Locations (1):
- Department of Anaesthesiology, University Hospital Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weiser TG, Haynes AB, Molina G, Lipsitz SR, Esquivel MM, Uribe-Leitz T, Fu R, Azad T, Chao TE, Berry WR, Gawande AA. Estimate of the global volume of surgery in 2012: an assessment supporting improved health outcomes. Lancet. 2015 Apr 27;385 Suppl 2:S11. doi: 10.1016/S0140-6736(15)60806-6. Epub 2015 Apr 26. PMID 26313057
- [Background] Weiser TG, Haynes AB, Molina G, Lipsitz SR, Esquivel MM, Uribe-Leitz T, Fu R, Azad T, Chao TE, Berry WR, Gawande AA. Size and distribution of the global volume of surgery in 2012. Bull World Health Organ. 2016 Mar 1;94(3):201-209F. doi: 10.2471/BLT.15.159293. PMID 26966331
- [Background] Berwanger O, Le Manach Y, Suzumura EA, Biccard B, Srinathan SK, Szczeklik W, Santo JA, Santucci E, Cavalcanti AB, Archbold RA, Devereaux PJ; VISION Investigators. Association between pre-operative statin use and major cardiovascular complications among patients undergoing non-cardiac surgery: the VISION study. Eur Heart J. 2016 Jan 7;37(2):177-85. doi: 10.1093/eurheartj/ehv456. Epub 2015 Sep 1. PMID 26330424
- [Background] Botto F, Alonso-Coello P, Chan MT, Villar JC, Xavier D, Srinathan S, Guyatt G, Cruz P, Graham M, Wang CY, Berwanger O, Pearse RM, Biccard BM, Abraham V, Malaga G, Hillis GS, Rodseth RN, Cook D, Polanczyk CA, Szczeklik W, Sessler DI, Sheth T, Ackland GL, Leuwer M, Garg AX, Lemanach Y, Pettit S, Heels-Ansdell D, Luratibuse G, Walsh M, Sapsford R, Schunemann HJ, Kurz A, Thomas S, Mrkobrada M, Thabane L, Gerstein H, Paniagua P, Nagele P, Raina P, Yusuf S, Devereaux PJ, Devereaux PJ, Sessler DI, Walsh M, Guyatt G, McQueen MJ, Bhandari M, Cook D, Bosch J, Buckley N, Yusuf S, Chow CK, Hillis GS, Halliwell R, Li S, Lee VW, Mooney J, Polanczyk CA, Furtado MV, Berwanger O, Suzumura E, Santucci E, Leite K, Santo JA, Jardim CA, Cavalcanti AB, Guimaraes HP, Jacka MJ, Graham M, McAlister F, McMurtry S, Townsend D, Pannu N, Bagshaw S, Bessissow A, Bhandari M, Duceppe E, Eikelboom J, Ganame J, Hankinson J, Hill S, Jolly S, Lamy A, Ling E, Magloire P, Pare G, Reddy D, Szalay D, Tittley J, Weitz J, Whitlock R, Darvish-Kazim S, Debeer J, Kavsak P, Kearon C, Mizera R, O'Donnell M, McQueen M, Pinthus J, Ribas S, Simunovic M, Tandon V, Vanhelder T, Winemaker M, Gerstein H, McDonald S, O'Bryne P, Patel A, Paul J, Punthakee Z, Raymer K, Salehian O, Spencer F, Walter S, Worster A, Adili A, Clase C, Cook D, Crowther M, Douketis J, Gangji A, Jackson P, Lim W, Lovrics P, Mazzadi S, Orovan W, Rudkowski J, Soth M, Tiboni M, Acedillo R, Garg A, Hildebrand A, Lam N, Macneil D, Mrkobrada M, Roshanov PS, Srinathan SK, Ramsey C, John PS, Thorlacius L, Siddiqui FS, Grocott HP, McKay A, Lee TW, Amadeo R, Funk D, McDonald H, Zacharias J, Villar JC, Cortes OL, Chaparro MS, Vasquez S, Castaneda A, Ferreira S, Coriat P, Monneret D, Goarin JP, Esteve CI, Royer C, Daas G, Chan MT, Choi GY, Gin T, Lit LC, Xavier D, Sigamani A, Faruqui A, Dhanpal R, Almeida S, Cherian J, Furruqh S, Abraham V, Afzal L, George P, Mala S, Schunemann H, Muti P, Vizza E, Wang CY, Ong GS, Mansor M, Tan AS, Shariffuddin II, Vasanthan V, Hashim NH, Undok AW, Ki U, Lai HY, Ahmad WA, Razack AH, Malaga G, Valderrama-Victoria V, Loza-Herrera JD, De Los Angeles Lazo M, Rotta-Rotta A, Szczeklik W, Sokolowska B, Musial J, Gorka J, Iwaszczuk P, Kozka M, Chwala M, Raczek M, Mrowiecki T, Kaczmarek B, Biccard B, Cassimjee H, Gopalan D, Kisten T, Mugabi A, Naidoo P, Naidoo R, Rodseth R, Skinner D, Torborg A, Paniagua P, Urrutia G, Maestre ML, Santalo M, Gonzalez R, Font A, Martinez C, Pelaez X, De Antonio M, Villamor JM, Garcia JA, Ferre MJ, Popova E, Alonso-Coello P, Garutti I, Cruz P, Fernandez C, Palencia M, Diaz S, Del Castillo T, Varela A, de Miguel A, Munoz M, Pineiro P, Cusati G, Del Barrio M, Membrillo MJ, Orozco D, Reyes F, Sapsford RJ, Barth J, Scott J, Hall A, Howell S, Lobley M, Woods J, Howard S, Fletcher J, Dewhirst N, Williams C, Rushton A, Welters I, Leuwer M, Pearse R, Ackland G, Khan A, Niebrzegowska E, Benton S, Wragg A, Archbold A, Smith A, McAlees E, Ramballi C, Macdonald N, Januszewska M, Stephens R, Reyes A, Paredes LG, Sultan P, Cain D, Whittle J, Del Arroyo AG, Sessler DI, Kurz A, Sun Z, Finnegan PS, Egan C, Honar H, Shahinyan A, Panjasawatwong K, Fu AY, Wang S, Reineks E, Nagele P, Blood J, Kalin M, Gibson D, Wildes T; Vascular events In noncardiac Surgery patIents cOhort evaluatioN (VISION) Writing Group, on behalf of The Vascular events In noncardiac Surgery patIents cOhort evaluatioN (VISION) Investigators; Appendix 1. The Vascular events In noncardiac Surgery patIents cOhort evaluatioN (VISION) Study Investigators Writing Group; Appendix 2. The Vascular events In noncardiac Surgery patIents cOhort evaluatioN Operations Committee; Vascular events In noncardiac Surgery patIents cOhort evaluatioN VISION Study Investigators. Myocardial injury after noncardiac surgery: a large, international, prospective cohort study establishing diagnostic criteria, characteristics, predictors, and 30-day outcomes. Anesthesiology. 2014 Mar;120(3):564-78. doi: 10.1097/ALN.0000000000000113. PMID 24534856
- [Background] Gillmann HJ, Meinders A, Grohennig A, Larmann J, Bunte C, Calmer S, Sahlmann B, Rustum S, Aper T, Lichtinghagen R, Koch A, Teebken OE, Theilmeier G. Perioperative levels and changes of high-sensitivity troponin T are associated with cardiovascular events in vascular surgery patients. Crit Care Med. 2014 Jun;42(6):1498-506. doi: 10.1097/CCM.0000000000000249. PMID 24584063
- [Background] Gillmann HJ, Meinders A, Larmann J, Sahlmann B, Schrimpf C, Aper T, Lichtinghagen R, Teebken OE, Theilmeier G. Adrenomedullin Is Associated With Surgical Trauma and Impaired Renal Function in Vascular Surgery Patients. J Intensive Care Med. 2019 Jan;34(1):67-76. doi: 10.1177/0885066616689554. Epub 2017 Jan 23. PMID 28110613
- [Background] International Surgical Outcomes Study group. Global patient outcomes after elective surgery: prospective cohort study in 27 low-, middle- and high-income countries. Br J Anaesth. 2016 Oct 31;117(5):601-609. doi: 10.1093/bja/aew316. PMID 27799174
- [Background] Devereaux PJ, Sessler DI. Cardiac Complications in Patients Undergoing Major Noncardiac Surgery. N Engl J Med. 2015 Dec 3;373(23):2258-69. doi: 10.1056/NEJMra1502824. No abstract available. PMID 26630144
- [Background] Antithrombotic Trialists' (ATT) Collaboration; Baigent C, Blackwell L, Collins R, Emberson J, Godwin J, Peto R, Buring J, Hennekens C, Kearney P, Meade T, Patrono C, Roncaglioni MC, Zanchetti A. Aspirin in the primary and secondary prevention of vascular disease: collaborative meta-analysis of individual participant data from randomised trials. Lancet. 2009 May 30;373(9678):1849-60. doi: 10.1016/S0140-6736(09)60503-1. PMID 19482214
- [Background] Bibbins-Domingo K; U.S. Preventive Services Task Force. Aspirin Use for the Primary Prevention of Cardiovascular Disease and Colorectal Cancer: U.S. Preventive Services Task Force Recommendation Statement. Ann Intern Med. 2016 Jun 21;164(12):836-45. doi: 10.7326/M16-0577. Epub 2016 Apr 12. PMID 27064677
- [Background] Williams CD, Chan AT, Elman MR, Kristensen AH, Miser WF, Pignone MP, Stafford RS, McGregor JC. Aspirin use among adults in the U.S.: results of a national survey. Am J Prev Med. 2015 May;48(5):501-8. doi: 10.1016/j.amepre.2014.11.005. PMID 25891049
- [Background] Wang Z, Gao F, Men J, Ren J, Modi P, Wei M. Aspirin resistance in off-pump coronary artery bypass grafting. Eur J Cardiothorac Surg. 2012 Jan;41(1):108-12. doi: 10.1016/j.ejcts.2011.04.021. PMID 21636287
- [Background] Kempfert J, Anger K, Rastan A, Krabbes S, Lehmann S, Garbade J, Sauer M, Walther T, Dhein S, Mohr FW. Postoperative development of aspirin resistance following coronary artery bypass. Eur J Clin Invest. 2009 Sep;39(9):769-74. doi: 10.1111/j.1365-2362.2009.02175.x. PMID 19674078
- [Background] Webster SE, Payne DA, Jones CI, Hayes PD, Bell PR, Goodall AH, Naylor AR. Anti-platelet effect of aspirin is substantially reduced after administration of heparin during carotid endarterectomy. J Vasc Surg. 2004 Sep;40(3):463-8. doi: 10.1016/j.jvs.2004.06.022. PMID 15337874